CLINICAL TRIAL: NCT06045078
Title: Aromatherapy for Post-operative Anxiety and Pain After Primary Unilateral Total Knee Replacement: a Pilot Randomized Controlled Trial
Brief Title: Aromatherapy in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-1715
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Total Knee Replacement; Post-operative Nausea and Vomiting; Opioid Use; Anxiety; Depression; Post Operative Pain
MeSH Terms: conditions — Vomiting; Anxiety Disorders; Depression; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Research staff (i.e. research assistants, coordinators, etc.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lavender-Peppermint Aromatherapy Group (Experimental): This is the interventional group. Participants in this group will receive aromatherapy tabs in the scent of lavender-peppermint. Tabs will be worn on a badge for a total of 72 hours, and participants will replace the aroma tabs every 12 hours.
  Interventions: Other: Elequil Lavender-peppermint Aromatabs
- Almond-oil Aromatherapy Group (Placebo Comparator): This is the placebo group. Participants in this group will receive aromatherapy tabs in the scent of almond oil. Tabs will worn on a badge for a total of 72 hours, and participants will replace the aroma tabs every 12 hours.
  Interventions: Other: Elequil Almond-Oil Aromatabs

INTERVENTIONS:
Other: Elequil Lavender-peppermint Aromatabs — 100% pure essential oils Lavender-peppermint aromatabs purchased through Beekley Medical
  Arms: Lavender-Peppermint Aromatherapy Group
Other: Elequil Almond-Oil Aromatabs — 100% pure essential oils Almond-oil aromatabs purchased through Beekley Medical
  Arms: Almond-oil Aromatherapy Group

SUMMARY:
The purpose of this pilot randomized controlled trial is to investigate the effects of aromatherapy on postoperative anxiety and pain in total knee replacement patients. The primary research questions are:

Does Lavender-Peppermint Aromatherapy reduce post operative anxiety in patients after primary total knee replacement when compared to placebo?

Does Lavender-Peppermint Aromatherapy reduce post operative pain in patient after primary total knee replacement when compared to placebo?

Participants will be assigned to one of the following groups at random:

* Intervention: Aromatherapy with the lavender-peppermint scent
* Control: Aromatherapy with the almond oil scent

Participants will also be asked to complete pre- and post-operative questionnaires.

Researchers will compare both groups (intervention vs control) to see if aromatherapy reduces post-operative anxiety and/or pain.

DETAILED DESCRIPTION:
Preoperative depression, anxiety, and catastrophizing have all been linked to an increase in postoperative pain and opiate use. Although aromatherapy, specifically lavender, may lower anxiety, no placebo-controlled trial has been undertaken to establish Aromatherapy's therapeutic promise for anxiety after total knee replacement. Although peppermint has been demonstrated to reduce nausea and vomiting, it has not been tested in this population for post-operative nausea and vomiting (PONV). The purpose of this pilot randomized controlled study is to determine the effectiveness of Lavender-Peppermint in reducing post-operative anxiety and discomfort in patients following unilateral primary knee replacement surgery.

The primary research questions are:

Does Lavender-Peppermint Aromatherapy reduce post operative anxiety in patients after primary total knee replacement when compared to placebo?

Does Lavender-Peppermint Aromatherapy reduce post operative pain in patient after primary total knee replacement when compared to placebo?

Participants will be assigned to one of the following groups at random:

* Intervention: Aromatherapy in the lavender-peppermint scent
* Control: Aromatherapy in the almond oil scent

Participants will also be asked to complete pre- and post-operative questionnaires via the following surveys/questionnaires:

* State-Trait Anxiety Inventory Short Form
* PROMIS Anxiety v1.0 (short form 8a)
* PROMIS Depression v1.0 (short form 8a)
* PROMIS Pain Interference v1.1 (short form 6b)
* Pain Catastrophizing Scale
* Pain Rating Scale in Numeric Form
* Opioid Consumption
* Opioid Related Symptoms Distress Scale
* Adverse Events
* Aromatherapy Satisfaction Questionnaire
* Bang Blinding Index

Researchers will compare both groups (intervention vs control) to see if aromatherapy reduces post-operative anxiety and/or pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and ≤ 80
* Scheduled to undergo primary, unilateral knee replacement surgery
* Willing and able to provide informed consent
* Willing and able to complete follow-up procedures
* Intact olfactory function
* Score 19 or greater on the PROMIS Anxiety Shortform 8A

Exclusion Criteria:

* Score <19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a
* Current major anxiety or depression
* Currently taking medications to treat anxiety
* Impaired sense of smell
* History of chronic pain with opioid use for greater than 3 months
* History of Drug or Alcohol abuse
* History of fibromyalgia
* History of G6PD deficiency
* Plant or tree nut allergy
* Severe allergy to Opioids, NSAIDS or local anesthetics (such as anaphylaxis)
* Severe liver disease, renal insufficiency (with inability to take acetaminophen or NSAIDS)
* Non-English Speaking
* Surgery requiring a hospitalization of greater than 3 days
* Patient refusal
* Current cardiac fibrillation
* Chronic opioid user (>3 months)
* BMI ≥ 45
* Contraindication to neuraxial anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in Anxiety level before and each individual day after surgery. | Measured pre-operatively, in the post-anesthesia care unit (PACU), post-operative day (POD) 1, POD 2, POD 3, POD 7
  To assess the change in participants' anxiety level before and each individual day after surgery. Measured using the State Anxiety Inventory.
  State anxiety was scored on the following scale:
  1. = not at all
  2. = somewhat
  3. = moderately so
  4. = very much so
  Trait anxiety was scored on the following scale:
  1. almost never
  2. sometimes
  3. often
  4. almost always
  with 1 being the lowest score and 4 being the highest score.
Difference in anxiety level before and after surgery | Measured pre-operatively and on post-operative day (POD) 7
  To assess participants' preoperative (cumulative 7 days before surgery) and postoperative (cumulative 7 days after surgery) anxiety. Measured using the PROMIS anxiety short form 8a Version 1.0. Scored on the following scale:
  1. = never
  2. = rarely
  3. = sometimes
  4. = often
  5. = always with 1 being the lowest score and 5 being the highest scores.
The average pain score after surgery | Measured pre-operatively, in the post-anesthesia care unit (PACU), post-operative day (POD) 1, POD 2, POD 3, POD 7
  To assess the average pain score of participants after surgery. Measured using the numerical rating scale (NRS). Measured on a 11-point numeric scale from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Difference in depression level before and after surgery | Measured pre-operatively and on post-operative day (POD) 7
  To assess participants' post-operative emotional distress. Measured using the PROMIS depression short form 8a. Scored on the following scale:
  1. = never
  2. = rarely
  3. = sometimes
  4. = often
  5. = always with 1 being the lowest score and 5 being the highest scores.
Average score on pain catastrophizing | Measured pre-operatively, post-operative day (POD) 1, POD 2, POD 3, POD 7
  The Pain Catastrophizing Scale is made up of 13 phrases that describe various thoughts and sensations that people may have while they are in pain. The items are assessed on a 5-point scale and are grouped into three categories: rumination, magnification, and helplessness. Scored on the following scale:
  0 = Not at all
  1. = To a slight degree
  2. = To a moderate degree
  3. = To a great degree
  4. = All the time with 0 being the lowest and 4 being the highest score.
Average score on pain interference | Measured pre-operatively and on post-operative day (POD) 7
  The PROMIS Pain Interference instruments (adult) measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items probing sleep and enjoyment in life, though the item bank only contains one sleep item. The Pain Interference items utilize a 7-day recall period (items include the phrase "the past 7 days"). Scored on the following scale:
  1. = Not at all
  2. = A little bit
  3. = Somewhat
  4. = Quite a bit
  5. = Very much With 1 being the lowest and 5 being the highest
Average post-operative opioid consumption | Measured in the post-operative care unit (PACU), post-operative day (POD) 1, POD2, POD3, POD7
  Self-reported measure of medication, dosage, and time of opioid consumption
Presence of post-operative nausea | Measured at post-anesthesia care unit (PACU), post-operative day (POD) 1, POD 2, POD 3, POD 7
  To assess if participants experience post-operative nausea. Measured using the Opioid Related Symptom Distress Scale question: In the past 24 hours, I had nausea (yes/no).
Presence of post-operative vomiting | Measured at post-anesthesia care unit (PACU), post-operative day (POD) 1, POD 2, POD 3, POD 7
  To assess if participants experience post-operative vomiting. Measured using the Opioid Related Symptom Distress Scale question: In the past 24 hours, I had vomiting (yes/no).
Incidences of post-operative complications | Measured at post-anesthesia care unit (PACU) up to post operative day 7
  To assess the incidences of post-operative complications such as need for ICU admission, DVT/PE, MI, stroke.
  To be measured in the number of patients who reported adverse events.
To assess the severity of opioid-related symptom distress | Measured at post-anesthesia care unit (PACU), post-operative day (POD) 1, POD 2, POD 3, POD 7
  The Opioid-Related Symptom Distress Scale (ORSDS) is a scale that assesses three dimensions of symptom distress (frequency, severity, and bothersomeness) for 12 symptoms. The symptom-specific ORSDS is calculated by taking the average of the three symptom distress dimensions.
  Frequency will be assessed using a 4 point scale:
  1. rarely
  2. occasionally
  3. frequently
  4. almost constantly with 1 being the lowest and 4 being the highest.
  Severity is assessed using a 4 point scale:
  1. slight
  2. moderate
  3. severe
  4. very severe with 1 being the lowest and 4 being the highest.
  Bothersomeness is assessed using a 5 point scale:
  1. not at all
  2. a little bit
  3. somewhat
  4. quite a bit
  5. very much with 1 being the lowest and 5 being the highest.
To assess participants' satisfaction with the aromatherapy | Measured at post operative day 7
  Self-reported responses on a survey of 7-items to assess participants' level of satisfaction with the aromatherapy they received.
  Measured on the following scale:
  1. = Not satisfied
  2. = A little bit
  3. = Moderately
  4. = Quite a bit
  5. = Extremely satisfied with 1 being the lowest and 5 being the highest.
Aromatab Adherence | Measured on post operative day (POD) 1, POD2, POD3.
  Feasibility was assessed as adherence to aromatab protocol was assessed as yes/no for whether the patient wore each of the 6 aromatabs.
Hospital Length of Stay | Measured at discharge as number of hours elapsed between post anesthesia care unit entry and discharge time
  Hospital length of stay was measured as hours elapsed from post anesthesia care unit entry to discharge.
Bang Blinding Index | Measured on postoperative day 7
  The Bang Blinding Index ranges from -1 to 1, where index of 1 indicates all responses are correct and complete unblinding is inferred. Patients and Research Assistants were asked to guess whether the patient was given the intervention (Lavender-Peppermint) or Control (Almond Oil) Aromatherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna Umeh, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Consensus Conference on 'Follow-up of Breast Cancer Patients'. Ann Oncol. 1995;6 Suppl 2:69-70. No abstract available. PMID 8547203
- [Background] Hunter JA, Zoma AA, Scullion JE, Protheroe K, Young AB, Sturrock RD, Capell HA. The geometric knee replacement in polyarthritis. J Bone Joint Surg Br. 1982;64(1):95-8. doi: 10.1302/0301-620X.64B1.7068729.
- [Background] Franco L, Blanck TJ, Dugan K, Kline R, Shanmugam G, Galotti A, von Bergen Granell A, Wajda M. Both lavender fleur oil and unscented oil aromatherapy reduce preoperative anxiety in breast surgery patients: a randomized trial. J Clin Anesth. 2016 Sep;33:243-9. doi: 10.1016/j.jclinane.2016.02.032. Epub 2016 May 5. PMID 27555173
- [Background] Wojcik A, Bonk K, Muller WU, Obe G, Streffer C. Do DNA double-strand breaks induced by Alu I lead to development of novel aberrations in the second and third post-treatment mitoses? Radiat Res. 1996 Feb;145(2):119-27. PMID 8606920
- [Background] Cunha GR, Shannon JM, Vanderslice KD, Sekkingstad M, Robboy SJ. Autoradiographic analysis of nuclear estrogen binding sites during postnatal development of the genital tract of female mice. J Steroid Biochem. 1982 Sep;17(3):281-6. doi: 10.1016/0022-4731(82)90201-1. PMID 7132346
- [Background] Mohr C, Jensen C, Padden N, Besel JM, Brant JM. Peppermint Essential Oil for Nausea and Vomiting in Hospitalized Patients: Incorporating Holistic Patient Decision Making Into the Research Design. J Holist Nurs. 2021 Jun;39(2):126-134. doi: 10.1177/0898010120961579. Epub 2020 Sep 27. PMID 32985338
- [Background] Briggs P, Hawrylack H, Mooney R. Inhaled peppermint oil for postop nausea in patients undergoing cardiac surgery. Nursing. 2016 Jul;46(7):61-7. doi: 10.1097/01.NURSE.0000482882.38607.5c. PMID 27333231
- [Background] Haward LR. Some psychological aspects of pregnancy. 16. Midwives Chron. 1969 May;83(976):171-2. No abstract available. PMID 5192342
- [Background] Woodall DL, Birken GA, Williamson K, Lobe TE. Isolated fetal-neonatal abdominal ascites: a sign of intrauterine intussusception. J Pediatr Surg. 1987 Jun;22(6):506-7. doi: 10.1016/s0022-3468(87)80207-5. No abstract available. PMID 3612440
- [Background] Kim JT, Ren CJ, Fielding GA, Pitti A, Kasumi T, Wajda M, Lebovits A, Bekker A. Treatment with lavender aromatherapy in the post-anesthesia care unit reduces opioid requirements of morbidly obese patients undergoing laparoscopic adjustable gastric banding. Obes Surg. 2007 Jul;17(7):920-5. doi: 10.1007/s11695-007-9170-7. PMID 17894152
- [Background] Kim JT, Wajda M, Cuff G, Serota D, Schlame M, Axelrod DM, Guth AA, Bekker AY. Evaluation of aromatherapy in treating postoperative pain: pilot study. Pain Pract. 2006 Dec;6(4):273-7. doi: 10.1111/j.1533-2500.2006.00095.x. PMID 17129308
- [Background] Soltani R, Soheilipour S, Hajhashemi V, Asghari G, Bagheri M, Molavi M. Evaluation of the effect of aromatherapy with lavender essential oil on post-tonsillectomy pain in pediatric patients: a randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1579-81. doi: 10.1016/j.ijporl.2013.07.014. Epub 2013 Aug 8. PMID 23932834
- [Background] Heidari Gorji MA, Ashrastaghi OG, Habibi V, Charati JY, Ebrahimzadeh MA, Ayasi M. The effectiveness of lavender essence on strernotomy related pain intensity after coronary artery bypass grafting. Adv Biomed Res. 2015 Jun 4;4:127. doi: 10.4103/2277-9175.158050. eCollection 2015. PMID 26261829
- [Background] Nasiri A, Mahmodi MA, Nobakht Z. Effect of aromatherapy massage with lavender essential oil on pain in patients with osteoarthritis of the knee: A randomized controlled clinical trial. Complement Ther Clin Pract. 2016 Nov;25:75-80. doi: 10.1016/j.ctcp.2016.08.002. Epub 2016 Aug 3. PMID 27863613
- [Background] Moeini M, Khadibi M, Bekhradi R, Mahmoudian SA, Nazari F. Effect of aromatherapy on the quality of sleep in ischemic heart disease patients hospitalized in intensive care units of heart hospitals of the Isfahan University of Medical Sciences. Iran J Nurs Midwifery Res. 2010 Fall;15(4):234-9. PMID 22049287
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Recklitis CJ, Blackmon JE, Chevalier LL, Chang G. Validating the Patient-Reported Outcomes Measurement Information System Short Form v1.0-Anxiety 8a in a sample of young adult cancer survivors: Comparison with a structured clinical diagnostic interview. Cancer. 2021 Oct 1;127(19):3691-3697. doi: 10.1002/cncr.33683. Epub 2021 Jul 1. PMID 34196978
- [Background] Karanika-Kouma A, Trigonidis G. [Pulpal reaction after the use of a glass ionomer cement as a cavity liner. An experimental study]. Hell Stomatol Chron. 1987 Jul-Sep;31(3):199-203. No abstract available. Greek, Modern. PMID 3153635
- [Background] Clover K, Lambert SD, Oldmeadow C, Britton B, Mitchell AJ, Carter G, King MT. Convergent and criterion validity of PROMIS anxiety measures relative to six legacy measures and a structured diagnostic interview for anxiety in cancer patients. J Patient Rep Outcomes. 2022 Jul 20;6(1):80. doi: 10.1186/s41687-022-00477-4. PMID 35857151